CLINICAL TRIAL: NCT00832117
Title: Phase 1 Study of Ixabepilone in Combination With Cisplatin in Subjects With Advanced Solid Tumors
Brief Title: Phase I Combination Ixabepilone + Cisplatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA163-177; 2008-004909-34
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Results first posted 2012-03-27 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — ixabepilone; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Escalation and Expansion (Experimental)
  Interventions: Drug: Ixabepilone; Drug: Cisplatin

INTERVENTIONS:
Drug: Ixabepilone — Escalation: Solution, intravenous (IV), 32-40 mg/m2, every 3 weeks, approximately 6 months
  Other Names: IXEMPRA®
Drug: Cisplatin — Escalation: Solution, IV, 60-100 mg/m2, every 3 weeks, approximately 6 months
Drug: Ixabepilone — Expansion: Solution, IV, 32 mg/m2, every 3 weeks, approximately 6 months
  Other Names: IXEMPRA®
Drug: Cisplatin — Expansion: Solution, IV, 60-80 mg/m2, every 3 weeks, approximately 6 months

SUMMARY:
The purpose of this study is to determine the highest dose of ixabepilone that can be given safely with cisplatin without causing severe or life-threatening side effects and for some patients with non-small cell lung cancer, the effects (good or bad) on your cancer will also be studied

ELIGIBILITY:
Escalation Phase Subjects: Primary solid tumor not curable by local measures such as surgery, radiation

Inclusion Criteria:

* Men and women age ≥ 18

Exclusion:

* More than 2 prior chemotherapy containing regimens for metastatic disease
* No prior exposure to cisplatin or ixabepilone

Expansion Phase Subjects: Advanced Non-small cell lung cancer

Inclusion Criteria:

* Men and women age ≥ 18

Exclusion:

* No prior chemotherapy-containing regimen for metastatic disease
* No prior exposure to cisplatin or ixabepilone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (7):
- United States (3):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - The Cancer Institute Of New Jersey, New Brunswick, New Jersey
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
- Italy (4):
  - Local Institution, Lucca
  - Local Institution, Meldola (Fc)
  - Local Institution, Rimini
  - Local Institution, Viterbo

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 30 participants were enrolled; 29 were treated (1 participant no longer met study criteria).
Groups:
- All Enrolled Participants: Participants received both ixabepilone (ixa) 32 mg/m^2+ cisplatin (cis) 60 mg/m^2 and ixa 32mg/m^2+cis 80mg/m^2, administered intravenously on Day 1 of a 21 day cycle.
Period: Overall Study
Arm/Group | All Enrolled Participants
Started | 29
Completed | 17
Not Completed | 12
Not completed — Death | 1
Not completed — Disease Progression | 11

BASELINE CHARACTERISTICS:
Groups:
- Ixa 32 mg/m^2+Cis 60 mg/m^2: 6 participants with solid tumors (refractory to prior therapy) in the dose-escalation phase and 18 participants (with no prior chemotherapeutic treatment) with NSCLC in the dose-expansion phase received ixabepilone (ixa) 32 mg/m^2+ cisplatin (cis) 60 mg/m^2 administered intravenously on Day 1 of a 21 day cycle
- 32mg/m^2+Cis 80mg/m^2: 5 participants in the dose-escalation phase with solid tumors (refractory to prior therapy) received ixa 32mg/m^2+cis 80mg/m^2, administered intravenously on Day 1 of a 21 day cycle
- Total: Total of all reporting groups
Arm/Group | Ixa 32 mg/m^2+Cis 60 mg/m^2 | 32mg/m^2+Cis 80mg/m^2 | Total
Number analyzed (Participants) | 24 | 5 | 29
Age, Continuous [Median (Full Range); unit: years] | 64 [33 to 77] | 54 [30 to 61] | 63 [30 to 77]
Age, Customized [Number; unit: participants]
  < 65 years | 12 | 5 | 17
  >= 65 years | 12 | 0 | 12
  < 50 years | 3 | 2 | 5
  >= 50 years | 21 | 3 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 12
  Male | 14 | 3 | 17
Karnofsky Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0-100, the lower the score, the worse the survival for most serious illnesses.
  participants
    80 - Activity with effort; some signs of disease | 9 | 2 | 11
    90 - Normal activity; minor signs of disease | 2 | 1 | 3
    100 - Normal no complaints; no evidence of disease | 13 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Participants Experiencing Dose Limiting Toxicity (DLT)
Description: DLT=any of the following treatment-related events:Grade(Gr)3/4 diarrhea despite the use of adequate/maximal medical intervention and/or prophylaxis;other Gr3 or greater nonhematological toxicity requiring removal from further study therapy;delayed recovery from treatment-related toxicity delaying scheduled retreatment for >3 weeks;Gr4 neutropenia (absolute neutrophil count <500 cells/mm^3) for >=5 consecutive days or Gr3/4 neutropenia of any duration with sepsis or fever >38.5°C;thrombocytopenia <25,000 cells/mm^3 or bleeding requiring platelet transfusion. Grades defined in Outcome Measure 7.
Time Frame: Within the first 21 days of first cycle
Population: all treated participants
Measure: Number; unit: participants
Arm/Group | Ixa 32 mg/m^2+Cis 60 mg/m^2 | 32mg/m^2+Cis 80mg/m^2
Number analyzed (Participants) | 24 | 5
participants | 0 | 2

2. Secondary Outcome: Number of Participants With Best Response As Assessed With Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Complete Response(CR):Disappearance of all clinical/radiological evidence of target lesions (TL) & all nontarget lesions (NTL) + no new lesions (NWL). Partial Response(PR):CR of TL + persistence of >=1 NTL (NonCR/NonPD) + no NWL; OR >=30% decrease in sum of longest diameter(LD) of all TL + CR or NonCR/NonPD in NTL + no NWL. Progressive Disease (PD):>=20% increase in sum of LD of TL regardless of NTL & NWL status; or unequivocal progression of NTL regardless of TL & NWL status; or NWL regardless of TL & NTL status. Stable Disease(SD): Neither PD nor PR in TL + CR or NonCR/NonPD in NTL + no NWL.
Time Frame: At End-of-Treatment visit. Median time on study therapy was 18 weeks (range: 6-69 weeks) for ixa 32 mg/m^2+cis 60 mg/m^2 arm; 6 weeks (range: 3-18 weeks) for ixa 32mg/m^2+cis 80 mg/m^2 arm.
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Ixa 32 mg/m^2+Cis 60 mg/m^2 | 32mg/m^2+Cis 80mg/m^2
Number analyzed (Participants) | 24 | 5
participants
  Complete Response | 0 | 0
  Partial Response | 8 | 0
  Stable Disease | 10 | 2
  Disease Progression | 5 | 2
  Not Assessed | 1 | 1

3. Primary Outcome: Maximum Tolerated Dose (MTD) and the Recommended Phase 2 Dose (RP2D) of Cisplatin in Combination With Ixabepilone, 32 mg/m^2
Description: The MTD is defined as the highest dose level in which dose limiting toxicities (DLTs) during the first 21 days of the first treatment cycle are observed in less than 1 out of 3 or less than 2 out of 6 treated subjects with at least 2 subjects experiencing DLT at the next higher dose level.
Time Frame: Within the first 21 days of first cycle
Population: All subjects who received at least 1 dose of either ixabepilone or carboplatin
Measure: Number; unit: mg/m^2
Groups:
- All Treated Participants: All participants who received at least 1 dose of either ixabepilone or carboplatin
Arm/Group | All Treated Participants
Number analyzed (Participants) | 29
mg/m^2 | 60

4. Secondary Outcome: Percentage of Participants With Response
Description: Response in participants with non-small cell lung cancer (NSCLC) was defined as the number of subjects in whose best response is partial response (PR) or complete response (CR) (see Outcome Measure 3 for definitions) divided by the total number of response evaluable subjects.
Time Frame: as for outcome 2
Population: This outcome measure was not analyzed as the indication for NSCLC is no longer being pursued.
Arm/Group | Ixa 32 mg/m^2+Cis 60 mg/m^2 | 32mg/m^2+Cis 80mg/m^2
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Duration of Response in Participants With Non-small Cell Lung Cancer (NSCLC)
Description: The duration of response will be computed for all treated subjects whose best response is either partial response (PR) or complete response (CR). The duration of response is measured from the time (in months) measurement criteria are first met for PR or CR, whichever is recorded first, until the date of documented progressive disease or death. Subjects who neither relapse nor die will be censored on the date of their last tumor assessment.
Time Frame: The duration of response is measured from the time (in months) measurement criteria are first met for PR or CR, whichever is recorded first, until the date of documented progressive disease or death. (Duration of study was approximately 21 months.)
Population: This outcome measure was not analyzed as the indication for NSCLC is no longer being pursued.
Arm/Group | Ixa 32 mg/m^2+Cis 60 mg/m^2 | 32mg/m^2+Cis 80mg/m^2
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious AEs (SAEs), Deaths, and Discontinuations Per National Cancer Institute (NCI) Common Terminology Criteria Adverse Events (CTCAE)Version 3 Criteria
Description: AE=any new untoward medical occurrence/worsening of a preexisting medical condition that does not necessarily have a causal relationship with treatment. SAE=any untoward medical event that results in death, persistent/significant incapacity, drug dependency or abuse; is life-threatening, an important medical event, a congenital anomaly/birth defect; requires/prolongs inpatient hospitalization. Treatment related=possibly, probably, or certainly related to and of unknown relationship to study treatment. Grade 1=Mild, 2=Moderate, 3=Severe/medically significant, 4=Life-threatening.
Time Frame: Assessed from the date of first dose until at least 30 days after the last dose of study drug. Median time on study therapy was 18 weeks (range: 6-69 weeks) for ixa 32 mg/m^2+cis 60 mg/m^2 arm; 6 weeks (range: 3-18 weeks) for ixa 32mg/m^2+cis 80 mg/m^2.
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Ixa 32 mg/m^2+Cis 60 mg/m^2 | 32mg/m^2+Cis 80mg/m^2
Number analyzed (Participants) | 24 | 5
participants
  Death | 4 | 1
  SAEs | 7 | 2
  Drug-Related SAEs | 4 | 1
  AEs Leading to Discontinuation | 2 | 0
  Drug-Related AEs Leading to Discontinuation | 1 | 0
  Overall AEs | 24 | 5
  Grade 3/4 AEs | 14 | 3
  Drug-Related AEs | 24 | 5
  Grade 3/4 Drug-Related AEs | 11 | 3

7. Secondary Outcome: Number of Participants With Laboratory Abnormalities Per National Cancer Institute (NCI) Common Terminology Criteria Adverse Events (CTCAE)Version 3 Criteria
Description: Grade (Gr) 1=Mild, 2=Moderate, 3=Severe/medically significant, 4=Life-threatening. Hemoglobin Gr1 <LLN - 10.0 g/dL; Gr2 <10.0 - 8.0 g/dL; Gr3 <8.0 - 6.5 g/dL; Gr4 <6.5 g/dL. White Blood Cell Count (WBC) Gr1 <lower limit of normal (LLN) - 3000/mm^3; Gr2 <3000 - 2000/mm^3; Gr3 <2000 - 1000/mm^3; Gr4 <1000/mm^3. Absolute Neutrophil Count (ANC) Gr 1 <LLN - 1500/mm^3; Gr 2 <1500 - 1000/mm^3; Gr3 <1000 - 500/mm^3; Gr 4 <500/mm^3. Platelets Gr1 <LLN - 75,000/mm^3; Gr2 <75,000 - 50,000/mm^3; Gr3 <50,000 - 25,000/mm^3; Gr4 <25,000/mm^3. Normal ranges vary by local laboratory.
Time Frame: Assessed at screening and weekly during treatment. Median time on study therapy was 18 weeks (range: 6-69 weeks) for ixa 32 mg/m^2+cis 60 mg/m^2 arm; 6 weeks (range: 3-18 weeks) for ixa 32mg/m^2+cis 80 mg/m^2.
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Ixa 32 mg/m^2+Cis 60 mg/m^2 | 32mg/m^2+Cis 80mg/m^2
Number analyzed (Participants) | 24 | 5
participants
  WBC, Grade 1-4 | 19 | 5
  WBC, Grade 3-4 | 6 | 3
  ANC, Grade 1-4 | 18 | 5
  ANC, Grade 3-4 | 12 | 4
  Platelet Count, Grade 1-4 | 9 | 3
  Platelet Count, Grade 3-4 | 0 | 1
  Hemoglobin, Grade 1-4 | 22 | 5
  Hemoglobin, Grade 3-4 | 1 | 0

ADVERSE EVENTS:
Groups:
- Ixa 32 mg/m2 + Cis 60 mg/m2: 6 participants with solid tumor (refractory to prior therapy) in the dose-escalation phase and 18 participants (with no prior chemotherapeutic treatment) for NSCLC in the dose-expansion phase received ixabepilone (ixa) 32 mg/m^2+ cisplatin (cis) 60 mg/m^2 administered intravenously on Day 1 of a 21 day cycle
- Ixa 32 mg/m2 +Cis 80 mg/m2: 5 participants in the dose-escalation phase with solid tumors (refractory to prior therapy) received ixa 32mg/m^2+cis 80mg/m^2, administered intravenously on Day 1 of a 21 day cycle
Arm/Group | Ixa 32 mg/m2 + Cis 60 mg/m2 | Ixa 32 mg/m2 +Cis 80 mg/m2
Serious Adverse Events (participants affected / at risk) | 7/24 | 2/5
Other Adverse Events (participants affected / at risk) | 24/24 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixa 32 mg/m2 + Cis 60 mg/m2 (N=24) | Ixa 32 mg/m2 +Cis 80 mg/m2 (N=5)
BACTERAEMIA (Infections and infestations) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
CEREBRAL ISCHAEMIA (Nervous system disorders) | 1 | 0
NEUTROPENIC SEPSIS (Infections and infestations) | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixa 32 mg/m2 + Cis 60 mg/m2 (N=24) | Ixa 32 mg/m2 +Cis 80 mg/m2 (N=5)
EAR PRURITUS (Ear and labyrinth disorders) | 0 | 1
MUCOSAL INFLAMMATION (General disorders) | 3 | 0
NAUSEA (Gastrointestinal disorders) | 16 | 3
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 0
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY MONILIASIS (Infections and infestations) | 0 | 1
TYMPANOMETRY ABNORMAL (Investigations) | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 1
DEPRESSION (Psychiatric disorders) | 0 | 2
DIZZINESS (Nervous system disorders) | 2 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 1
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 0
PLATELET COUNT DECREASED (Investigations) | 1 | 1
PYREXIA (General disorders) | 3 | 1
ANXIETY (Psychiatric disorders) | 1 | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 3 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 8 | 2
OEDEMA PERIPHERAL (General disorders) | 3 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
TACHYCARDIA (Cardiac disorders) | 2 | 1
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 1
HEADACHE (Nervous system disorders) | 2 | 1
HYPERMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 3 | 1
OEDEMA (General disorders) | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 1
WEIGHT DECREASED (Investigations) | 2 | 0
ANAEMIA (Blood and lymphatic system disorders) | 4 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 2
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 0 | 1
PAIN (General disorders) | 3 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 8 | 3
ASTHENIA (General disorders) | 5 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 6 | 0
DYSGEUSIA (Nervous system disorders) | 5 | 1
EAR PAIN (Ear and labyrinth disorders) | 0 | 1
FLUSHING (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0
NEUROTOXICITY (Nervous system disorders) | 4 | 0
RASH (Skin and subcutaneous tissue disorders) | 3 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 1
BLOOD CREATININE INCREASED (Investigations) | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2 | 0
HERPES VIRUS INFECTION (Infections and infestations) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1
NEUTROPHIL COUNT DECREASED (Investigations) | 1 | 2
CONSTIPATION (Gastrointestinal disorders) | 7 | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 | 0
EAR CANAL ERYTHEMA (Ear and labyrinth disorders) | 0 | 1
FATIGUE (General disorders) | 10 | 4
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 2
VOMITING (Gastrointestinal disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.